CLINICAL TRIAL: NCT01027442
Title: Conventional Versus Computer Aided Implantology
Brief Title: The Use of Bone-, Tooth- and Mucosa- Supported Stereolithographic Guides for Dental Implant Placement
Acronym: stereolitho
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: Risus medikal, Thommen medical (Switzerland) Turkish partner (Unknown); Dentsply Implants Manufacturing GmbH (Industry)
Responsible Party: Istanbul University, Faculty of Dentistry
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Stereolithographic guides; Implant with SLA (Other: Istanbul University, Faculty of Dentistry)
Record Dates: First submitted 2009-12-07; First posted 2009-12-08 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2007-06

CONDITIONS: Stereolithography; Dental Implants; Prosthesis
Keywords: Stereolithography; Dental implants,; Prosthetics; positioning-errors; logistic regression analysis
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional implant placement method (Placebo Comparator): The patients in ths group will be treated by conventional, "free-hand" implant placement
  Interventions: Device: Dental Implants
- Computer-guidedimplant placement (Active Comparator): In this group, the patients will be treated by implants placed via computer generated SLA guides
  Interventions: Device: Mucosa-supported single-type guides; Device: Bone-supported guides

INTERVENTIONS:
Device: Mucosa-supported single-type guides — Compute generated Mucosa-supported single-type guides
  Other Names: Simplant, SAFEsystem, Materialise Dental, Leuven , Belgium
  Arms: Computer-guidedimplant placement
Device: Bone-supported guides — Computer generated, Multiple type Bone-supported guides
  Other Names: Aytasarim, Classic. Odtu-Kosgep, Ankara, Turkey
  Arms: Computer-guidedimplant placement
Device: Dental Implants — Dental implants placed via conventional free-hand method
  Other Names: Thommen Medical SPI, Waldenburg, Switzerland; Frident Xixe, dentsply Friadent-Turkey
  Arms: Conventional implant placement method

SUMMARY:
Introduction:

The use stereolithographic (SLA) guides may provide significant benefits in simultaneous placement of multiple implants, especially in large edentulous areas lacking anatomic landmarks for surgical reference. Planning of the implant positions prior to surgery may shorten the duration of the surgery spent by exploring and determining the suitable implant location on the edentulous alveolar crest in the standard technique . Previous studies have demonstrated the use of many SLA guide in this manner, however; most were designed to be used as placed on the alveolar crest (bone-supported) following a flap exposure, and there was no depth-control of the osteotomy drills. Further advances in stereolithography allowed flapless surgeries to be performed via mucosa-supported guides (Rosenfeld, et al. 2006c, Tardieu, et al. 2007). The use of these guides eliminates not only the time required for incision and flap exposure but post-operative patient morbidity and discomfort may also be reduced, due to the non-invasive nature of the procedure. The aim of this study is to investigate the accuracy, surgical and post-operative complications and post-loading outcomes of implants placed by the conventional and aforementioned computer-aided methods.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patient with at leat one edentuşous jaw

Exclusion Criteria:

* Patients with at least one edentulous jaw with healthy systemic and oral status without severe alveolar bone athrophy, major alveolar hard and/or soft tissue deficiency, mouth opening restriction, heavy smoking (> 10 /per day) and parafunctional habits were included in the study.
* All patients were initially evaluated for the suitability of an implant supported fixed prosthesis and any patients unsuitable for such prosthetic superstructure (i.e. severe hard and soft tissue athrophy, insufficient hygiene practice etc.) were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-07; Primary Completion 2009-01 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tayfun Ozdemir, Prof.Dr., Study Chair — Section head: Department of Implantology, Faculty of Dentistry, Istabul University; Volkan Arısan, Dr.Med.Dent, Principal Investigator — Department of Oral Implantology, Istanbul University; Cuneyt Z Karabuda, Prof.Dr., Study Director — Department of Oral Implantology, Istanbul University
Locations (1):
- Department of Oral Implantology, Faculty of Dentistry, ıstnabul University, Istanbul, Capa, Turkey (Türkiye)

REFERENCES:
- [Result] Arisan V, Karabuda ZC, Ozdemir T. Accuracy of two stereolithographic guide systems for computer-aided implant placement: a computed tomography-based clinical comparative study. J Periodontol. 2010 Jan;81(1):43-51. doi: 10.1902/jop.2009.090348. PMID 20059416
- [Result] Arisan V, Karabuda CZ, Ozdemir T. Implant surgery using bone- and mucosa-supported stereolithographic guides in totally edentulous jaws: surgical and post-operative outcomes of computer-aided vs. standard techniques. Clin Oral Implants Res. 2010 Sep;21(9):980-8. doi: 10.1111/j.1600-0501.2010.01957.x. Epub 2010 May 24. PMID 20497439
- [Result] Arisan V, Karabuda CZ, Mumcu E, Ozdemir T. Implant positioning errors in freehand and computer-aided placement methods: a single-blind clinical comparative study. Int J Oral Maxillofac Implants. 2013 Jan-Feb;28(1):190-204. doi: 10.11607/jomi.2691. PMID 23377066
- [Result] Arisan V, Bolukbasi N, Oksuz L. Computer-assisted flapless implant placement reduces the incidence of surgery-related bacteremia. Clin Oral Investig. 2013 Dec;17(9):1985-93. doi: 10.1007/s00784-012-0886-y. Epub 2012 Dec 6. PMID 23224042